CLINICAL TRIAL: NCT02798848
Title: Tablet Computers Versus Optical Aids to Support Education and Learning in Children and Young People With Low Vision: a Pilot Randomized Controlled Trial
Brief Title: CREATE - Children Reading With Electronic Assistance To Educate
Acronym: CREATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: L.V. Prasad Eye Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 15/0570
Record Dates: First submitted 2016-04-19; First posted 2016-06-14 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-04

CONDITIONS: Vision, Low; Child; Adolescent Development
MeSH Terms: conditions — Vision, Low

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Assistive technology: tablet computer (Experimental): iPad tablet computers
  Interventions: Device: Tablet computer
- Standard optical low vision devices (Active Comparator): standard optical devices including magnifiers, telescopes, CCTV
  Interventions: Device: Tablet computer

INTERVENTIONS:
Device: Tablet computer — iPad

SUMMARY:
This pilot randomized controlled trial (RCT) will test the methodology for a full RCT of assistive technologies for children/young people with low vision/blindness. The investigators will recruit 40 students age 10-18 years in India and the UK, who will be randomised into two groups. Apple iPads will be the active intervention; the control arm will be the local standard low-vision aid care. Primary outcomes will be acceptance/usage and accessibility of the device and trial feasibility measures. Exploratory outcomes will be validated measures of vision-related quality of life for children/young people as well as validated measures of reading and educational outcomes. In addition, the investigators will carry out semistructured interviews with the participants and their teachers, and attempt to evaluate cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

* age 10-18 years
* low vision, defined as "best corrected visual acuity (BCVA) for distance between - less than 6/18 (0.48 logMAR) and 3/60 (1.30 logMAR) in the better eye" (WHO) ability to read printed material
* no previous or current use of a tablet computer for educational purposes We will include students who have access to a tablet computer already, but only use it for recreational purposes. We will also include students who use a laptop. We will also include students who use or have previously used optical low-vision aids such as magnifiers, telescopes and CCTV systems.

Exclusion Criteria:

* current or previous use of a tablet computer for educational purposes

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-12 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
acceptance/usage, measured as ordinal variable by participant diary | six months
  0 = no acceptance, 1 = acceptance as described, 2 = used frequently
accessibility measured as ordinal variable as score on a touch-based game, "Piano Tiles" | six months
  0 = not accessible,
  1 = accessible with help, 2 = accessible independently
recruitment rates into the trial | six months
  recruitment rate and reasons for not taking part

SECONDARY OUTCOMES:
Cardiff Visual Ability Questionnaire for Children (CVAQC) score | six months
  Functional visual ability scale, for participants in the UK
LV Prasad Functional Vision Questionnaire | six months
  Vision related quality of life scale, for participants in India
Impact of Vision Impairment for Children (IVI_C) Questionnaire | six months
  Functional vision, all participants
Neale Analysis of Reading Ability (NARA) | six months
  reading accuracy, comprehension and speed
International Reading Speed Texts (IREST) | six months
  reading speed

CONTACTS AND LOCATIONS:
Overall Officials: Annegret Dahlmann-Noor, PhD, Principal Investigator — Moorfields Eye Hospital NHS Foundation Trust
Locations (3):
- Meera and L B Deshpande Centre for Sight Enhancement, L V Prasad Eye Institute, Hyderabad, India
- United Kingdom (2):
  - South Essex Partnership Foundation Trust - Child Development Centre Bedford, Bedford
  - Moorfields Eye Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gothwal VK, Thomas R, Crossland M, Bharani S, Sharma S, Unwin H, Xing W, Khabra K, Dahlmann-Noor A. Randomized Trial of Tablet Computers for Education and Learning in Children and Young People with Low Vision. Optom Vis Sci. 2018 Sep;95(9):873-882. doi: 10.1097/OPX.0000000000001270. PMID 30153236
- [Derived] Crossland MD, Thomas R, Unwin H, Bharani S, Gothwal VK, Quartilho A, Bunce C, Dahlmann-Noor A. Tablet computers versus optical aids to support education and learning in children and young people with low vision: protocol for a pilot randomised controlled trial, CREATE (Children Reading with Electronic Assistance To Educate). BMJ Open. 2017 Jun 21;7(6):e015939. doi: 10.1136/bmjopen-2017-015939. PMID 28637740